CLINICAL TRIAL: NCT00201331
Title: Prospective Phase II Randomized Trial of Postoperative Adjuvant Chemotherapy in Patients With High Risk Colon Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Health Research Institutes, Taiwan (Other)
Collaborators: Chang Gung Memorial Hospital (Other); Changhua Christian Hospital (Other); China Medical University Hospital (Other); Mackay Memorial Hospital (Other); Chi Mei Medical Hospital (Other); Kaohsiung Veterans General Hospital. (Other); National Cheng-Kung University Hospital (Other); Taichung Veterans General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: T1202
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2005-12-16 (Estimated); Status verified 2005-12

CONDITIONS: Colonic Diseases; Adenocarcinoma
MeSH Terms: conditions — Colonic Diseases; Adenocarcinoma

INTERVENTIONS:
Drug: leucovorin+5-FU

SUMMARY:
Based on the astonishing high response rate in metastatic colorectal cancer in weekly high dose 5-FU and leucovorin, we will conduct a clinical trial to clarify the activity of this regimen in the adjuvant setting. The regimen of 5-FU and high dose leucovorin administered as the schedule of INT-0089 will be chosen as the controlled arm which was proven as effective as standard 5-FU plus levamisole regimen with short duration of treatment.21 In this study, continuous infusion of 5-FU (HDFL, Arm B) and bolus injection of 5-FU (Arm A) will be administered to the high risk colon cancer(N2 disease) patients. The role of TS level and inhibition of TS as a predictor of adjuvant chemotherapy with 5-FU based treatment will be clearly defined prospectively.

DETAILED DESCRIPTION:
Approximately 75% of all patients with colon carcinoma present at a stage when all gross tumor can be surgically resected. Despite that high resectability rate, about 50% of all colon adenocarcinoma patients die of subsequent metastatic disease not apparent at surgery. These individuals could benefit from adjuvant local or systemic chemotherapy.

Based on the encouraging antitumor activity of 5-FU plus leucovorin(LV) in patients with metastatic colon carcinoma6,7, several investigators reported their results using this combination in the adjuvant setting. Results of an NSABP C-038 suggested that postoperative 5-FU plus leucovorin reduces the risk of colon cancer recurrence by 30% and the associated mortality by 32% compared with MOF(semustine, vincristine, and 5-FU). Recently, investigators from the IMPACT group9 analyzed the role of adjuvant 5-FU plus high dose leucovorin given 5 days every 28 days for a total of six courses versus no treatment in patients with stage II or III colon cancer. The treatment arm showed a significant reduction (by 22%) in mortality (P=0.029) and a 35% reduction in relapse rate (P=0.0001). Preliminary results from other studies have also suggested benefits of 5-FU plus leucovorin as adjuvant treatment of colon cancer10,11,12. Those studies had employed chemotherapy with 5-FU plus leucovorin, although there were differences in duration of treatment and drug dose among those trials, it is striking that all revealed a similar magnitude of benefit for adjuvant chemotherapy with 5-FU and leucovorin in node positive patients. At the present time, both 5-FU plus levamisole and 5-FU plus leucovorin can be considered acceptable adjuvant chemotherapy regimens for patients with node positive disease.

Thymidylate synthase(TS) is a critical therapeutic target for the fluoropyrimidine cytotoxic drugs that are the mainstay of the treatment for patients with advanced colorectal cancer. TS provide the sole de nono source of thymidylate for DNA synthesis. The clinical importance of TS in determining fluoropyrimidine cytotoxicity has been established in both clinical and preclinical study. Increased expression of TS protein due to underlying gene amplification has been described in cell lines selected for drug resistance by exposure to 5-FU.22,23 Several investigators have also demonstrated that intratumoral TS activity are predictive for response to 5-FU.24-26 High TS activity was associated with no response, whereas a low TS activity was associated with good response to 5-FU.

ELIGIBILITY:
Inclusion Criteria:

Signed written informed consent. Curative resection of colon cancer and upper rectal cancer, which is not planned for radiotherapy. Histologically proved adenocarcinoma of the colon. Stages: T1-4N2M0 (LN ≧4) Age less or equal to 70 years old. Performance status: 0 to 1 (ECOG) Adequate liver function (Bil. < 2 mg/dl, GOT, GPT< 3x normal limit) Adequate renal function (Cr < 2.0 mg/dl) Adequate bone marrow function(WBC ≧3500/mm3, Platelet ≧100000/mm3) Individual regular follow-up possible. 3.320 Patient who can receive adjuvant chemotherapy within 6 weeks after operation.

Patient who can receive a "indwelling catheter" surgery.

Exclusion Criteria:

Uncontrolled intercurrent illness, e.g. active infection or concurrent major systemic disease (e.g. psychosis, ESRD, heart failure [NYHA class III], liver cirrhosis [Child B&C], or AIDS). Intestinal obstruction or occlusion postoperation. Pregnant or lactating woman. Allergy to 5-Fluorouracil or leucovorin. Other primary cancer except skin squamous or basal cell carcinoma or cured in-situ cancer of the cervix.

Previous treatment of chemotherapy or radiotherapy.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162
Dates: Start 2002-04; Study Completion 2012-10

PRIMARY OUTCOMES:
To compare the DFS and OS of HDFL vs. weekly bolus 5-FU plus high dose LV as adjuvant chemotherapy for N2 colon cancer

SECONDARY OUTCOMES:
1. To evaluate safety and toxicity of both arm
2. To assess the impact of TS overexpression on patients with resectable N2 colon carcinoma.
3. To assess the disease-free survival of patients with high or low TS level of N2 colon cancer, when adjuvant chemotherapy of 5-FU was administered by bolus or continuous infusion .

CONTACTS AND LOCATIONS:
Overall Officials: Cheng-Yi Wang, PHD, Study Chair — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan

REFERENCES:
- See also: Related Info — http://www.nhri.org.tw